CLINICAL TRIAL: NCT05179018
Title: Clinical and Diagnostic Value of Ribosomal p2 Autoantibodies in Systemic Lupus Erythematosus: Case Control Study
Brief Title: Clinical and Diagnostic Value of Ribosomal p2 Autoantibodies in Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna Allah Nashaat, Principal investigator, Assiut University
Other Study IDs: Rib P2 antibodies in sle pts
Record Dates: First submitted 2021-12-18; First posted 2022-01-05 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLE patients group: The study will include 50 patients suffering from SLE, all patients with SLE should fulfill 2012 SLICC criteria
  Interventions: Diagnostic Test: Ribosomal p2 Autoantibodies as a Serum marker
- Healthy control group: Control group of 40 healthy volunteers with age and gender-matched with SLE patients.
  Interventions: Diagnostic Test: Ribosomal p2 Autoantibodies as a Serum marker

INTERVENTIONS:
Diagnostic Test: Ribosomal p2 Autoantibodies as a Serum marker — Using serum marker

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disorder characterized by production of autoantibodies directed against nuclear and cytoplasmic antigens. Clinically, this disorder is characterized by periods of remission and relapse (1). The early and accurate diagnosis of SLE is challenging (2).

The SLE pathogenesis involves multiple cellular components of the innate and immune systems, presence of autoantibodies and immune complexes, engagement of the complement system and cytokine dysregulation (3). About 180 autoantibodies have been identified in SLE patients, 102 of which are reported to have an organ-specific correlation with SLE disease identified in SLE patients, with SLE disease activity (4). However, with the exception of autoantibodies such as antinuclear antibody (ANA), anti double stranded DNA (dsDNA), anti-smith and antiphospholipid antibodies, currently proposed by the American college of rheumatology (ACR) (5)

DETAILED DESCRIPTION:
systemic lupus international collaborating clinics (SLICC) (6) for the diagnosis of SLE, most of these autoantibodies lack sufficient sensitivity and/or specificity for use in clinical diagnosis. Discovery of additional autoantibodies with high sensitivity and specificity is important for early diagnosis and assessment of the prognosis of SLE (7).

Anti-ribosomal P(Anti-Rib-P) antibody, routinely tested in SLE, targets a homologous 22-amino acid C-terminal (C-22) sequence shared by three ribosomal phosphoproteins known as P0, P1, and P2 (8).

The prevalence of anti-Rib-P antibody is about 15-40% in SLE patients and varies with the ethnicity, disease activity and detection method (9). Studies have disclosed that anti-P antibodies react with activated T cells but not with B cells, suggesting possible direct effects of anti-P antibodies on immune regulation (10).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfilled the 2012 SLICC criteria (6).
2. SLE Patients >= 18 years old.

Exclusion Criteria:

* 1-SLE Patients < 18 years old. 2- Patients with other autoimmune diseases or malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SLE pts obtained from rheumatology clinic in assiut university hospital >= 18 years
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
a. Primary (main): Assessment of diagnostic value (sensitivity and specificity) of serum ribosomal p2 autoantibody level in SLE patients in comparison to healthy controls | Baseline
  The importance of Ribosomal p2 autoantibodies in diagnosis of SLE

SECONDARY OUTCOMES:
b. Secondary (subsidiary): correlation between serum ribosomal p2 autoantibody level and SLE clinical, laboratory data, disease activity and severity. | Baseline
  The relation between rib p2 level in serum and determination of disease severity and prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Samar Hassanein goma, MD, Study Director — Assiut university Egypt; Maha Sayed ibrahim, MD, Study Director — Assiut university Egypt

REFERENCES:
- [Background] Fortuna G, Brennan MT. Systemic lupus erythematosus: epidemiology, pathophysiology, manifestations, and management. Dent Clin North Am. 2013 Oct;57(4):631-55. doi: 10.1016/j.cden.2013.06.003. PMID 24034070
- [Background] Thong B, Olsen NJ. Systemic lupus erythematosus diagnosis and management. Rheumatology (Oxford). 2017 Apr 1;56(suppl_1):i3-i13. doi: 10.1093/rheumatology/kew401. PMID 28013206
- [Background] Fava A, Petri M. Systemic lupus erythematosus: Diagnosis and clinical management. J Autoimmun. 2019 Jan;96:1-13. doi: 10.1016/j.jaut.2018.11.001. Epub 2018 Nov 16. PMID 30448290
- [Background] Yaniv G, Twig G, Shor DB, Furer A, Sherer Y, Mozes O, Komisar O, Slonimsky E, Klang E, Lotan E, Welt M, Marai I, Shina A, Amital H, Shoenfeld Y. A volcanic explosion of autoantibodies in systemic lupus erythematosus: a diversity of 180 different antibodies found in SLE patients. Autoimmun Rev. 2015 Jan;14(1):75-9. doi: 10.1016/j.autrev.2014.10.003. PMID 25449682
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus. Ann Rheum Dis. 2019 Sep;78(9):1151-1159. doi: 10.1136/annrheumdis-2018-214819. Epub 2019 Aug 5. PMID 31383717
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Ling HZ, Xu SZ, Leng RX, Wu J, Pan HF, Fan YG, Wang B, Xia YR, Huang Q, Shuai ZW, Ye DQ. Discovery of new serum biomarker panels for systemic lupus erythematosus diagnosis. Rheumatology (Oxford). 2020 Jun 1;59(6):1416-1425. doi: 10.1093/rheumatology/kez634. PMID 31899518
- [Background] Mahler M, Kessenbrock K, Raats J, Williams R, Fritzler MJ, Bluthner M. Characterization of the human autoimmune response to the major C-terminal epitope of the ribosomal P proteins. J Mol Med (Berl). 2003 Mar;81(3):194-204. doi: 10.1007/s00109-003-0423-1. Epub 2003 Mar 14. PMID 12682728
- [Background] Mahler M, Kessenbrock K, Raats J, Fritzler MJ. Technical and clinical evaluation of anti-ribosomal P protein immunoassays. J Clin Lab Anal. 2004;18(4):215-23. doi: 10.1002/jcla.20026. PMID 15202113
- [Background] Nagai T, Arinuma Y, Yanagida T, Yamamoto K, Hirohata S. Anti-ribosomal P protein antibody in human systemic lupus erythematosus up-regulates the expression of proinflammatory cytokines by human peripheral blood monocytes. Arthritis Rheum. 2005 Mar;52(3):847-55. doi: 10.1002/art.20869. PMID 15751081
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Background] Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is valid, and renal and pulmonary organ scores are predictors of severe outcome in patients with systemic lupus erythematosus. Br J Rheumatol. 1996 Mar;35(3):248-54. doi: 10.1093/rheumatology/35.3.248. PMID 8620300